CLINICAL TRIAL: NCT03126903
Title: A Prospective, Multicenter Clinical Trial Designed to Evaluate the Safety and Probable Benefit of the KeraKlear Non-Penetrating Keratoprosthesis in Subjects With Corneal Opacity With Poor Prognosis for Corneal Transplant
Brief Title: A Clinical Study to Evaluate the KeraKlear Keratoprosthesis in Patients With Corneal Opacity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: KeraMed is being discontinued because it is no longer feasible due to the slow pace of recruitment and insufficient financial resources.
Sponsor: KeraMed, Inc. (Industry)
Collaborators: National Eye Institute (NEI) (NIH); ClinReg Consulting Services, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KERA002; 1R44EY021664-01 (NIH)
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Corneal Blindness

STUDY DESIGN:
Intervention Model Description: Single arm, open-label clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single-Arm (Experimental): KeraKlear Non-Penetrating Keratoprosthesis
  Interventions: Device: KeraKlear Non-Penetrating Keratoprosthesis

INTERVENTIONS:
Device: KeraKlear Non-Penetrating Keratoprosthesis — The KeraKlear is a flexible non-penetrating artificial cornea designed to be implanted through small corneal incisions in subjects with corneal opacity.

SUMMARY:
To evaluate the safety and probable benefit of the KeraKlear Non-Penetrating Keratoprosthesis when implanted in an eye with corneal opacity that is at high risk of complications with PK.

DETAILED DESCRIPTION:
To evaluate the safety and probable benefit of the KeraKlear Non-Penetrating Keratoprosthesis when implanted in an eye with corneal opacity that is at high risk of complications with PK. A prospective, multicenter, clinical trial, designed to demonstrate the safety and performance of the KeraKlear Non-Penetrating Keratoprosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Corneal blindness where cornea transplantation is necessary but with a high risk of graft failure due to

  1. severe limbal stem cell deficiency (LSCD) associated with aniridia or
  2. one full-thickness graft failure and at high risk of a failed second graft; specifically, those who have either young recipient age (age less than 40 years), a history of anterior segment surgery (in addition to prior PKP), and/or pre-operative glaucoma or
  3. multiple (two or more) failed cornea transplantation surgeries and spontaneous visual improvement without surgical intervention is not expected or probable.
* Best Corrected Distance Visual Acuity (Snellen) which is equal or worse than 20/200 in the study eye (but at least light perception with projection)
* Estimated visual potential of the study eye is greater than or equal to at least two lines visual improvement of BCDVA of current vision in the study eye.
* Patient and/or caregiver willing and able to insert and remove bandage contact lens.

Exclusion Criteria:

* Visual Acuity of No Light Perception (NLP) in the study eye
* The patient is monocular or the non-study eye has Best Corrected Distance Visual Acuity (Snellen) of worse than 20/160 due to an ocular condition other than severe aniridic limbal stem cell deficiency or failed cornea transplantation surgery(ies).
* Suitable for standard PK with donor tissue in the study eye.
* History of severe dry eye syndrome or a Schirmer test with results of less than 3mm after 5 minutes of testing with the use of topical anesthetic in either eye.
* Active or history of an auto-immune disease (e.g. Rheumatoid Arthritis, Ocular Cicatricial Pemphigoid, Lupus, Steven's Johnson Syndrome, atopic keratoconjunctivitis, etc.).
* On medications that may affect wound healing, such as antimetabolites or other chemotherapeutic agents.
* History of posterior segment eye disease in either eye (including macular degeneration, optic neuropathy, posterior uveitis) which is expected to limit the visual improvement to less than two lines of vision.
* History of retinal surgery in the fellow eye (including retinal detachment repair, intravitreal injection etc.).
* History of retinal surgery in the study eye (including retinal detachment repair, intravitreal injection, etc.) unless the vision is at least light perception with projection in four field quadrants and the macula is attached (if there is no view of the retina, an ultrasound must show the macula is attached).
* History of uncontrolled glaucoma in either eye (IOP has been measured above 25 mmHg at any time in the last 6 months).
* Current use of beta blocker eye drops (e.g. timolol, levobunolol, etc.).
* Vertical cup-to-disc (C:D) ratio greater than or equal to 0.8 in either eye (if able to visible through corneal opacity). If not visible, patient is not to be excluded.
* Limited visual potential (patient does not have the ability to improve a minimum of two lines of vision of BCDVA by history).
* History of amblyopia in the study eye limiting visual potential.
* If the patient has had a corneal transplant, corneal transplantation surgery was performed less than 2 years ago.
* Anticipated need for surgery on the study eye during the course of the study (including cataract surgery).
* Aphakia in the study eye.
* Active ocular infection in either eye.
* Hypotony in the study eye (IOP < 6mmHg).
* History of herpetic ocular infection in the study eye.
* Corneal thickness less than 400 microns in any region of the pachymetry map, i.e.

lamellar resection depth would be <100 microns from corneal endothelium accounting for the optic height of the selected implant design (i.e. 300 microns for KeraKlear or 500 microns for KeraKlear XT model).*.

* Inability to protect the operated eye from trauma.
* Females who are pregnant, lactating, or unwilling to use adequate birth control for t the duration of the study.
* Patient is currently taking Sumatriptan (Imitrex) and unable to discontinue during the study.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Improvement in BCDVA compared to baseline | Baseline, Month 1, Month 2, Month 3, Month 4, Month 6, Month 9 and Month 12
  Best Corrected Distance Visual Acuity (BCDVA) will be measured in the study eye. An ETDRS visual acuity chart will be used to measure BCDVA at baseline, Month 1, Month 2, Month 3, Month 4, Month 6, Month 9, and Month 12.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of California Irvine, Irvine, California
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - Massachussetts Eye and Ear Infirmary, Boston, Massachusetts
  - Duke University School of Medicine - Dept. of Ophthalmology, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kilian R, Lammer J, Roberts P, Rizzo C, Pedrotti E, Marchini G, Schmidinger G. Nonpenetrating Foldable Intrastromal Keratoprosthesis: A Review of the Literature. Cornea. 2024 Jul 1;43(7):909-915. doi: 10.1097/ICO.0000000000003500. Epub 2024 Feb 21. PMID 38381061